CLINICAL TRIAL: NCT05273606
Title: A Clinical Study of Short-term Clinical Performance of Multifocal Soft Contact Lens
Brief Title: Short-term Clinical Performance of Multifocal Soft Contact Lens
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiao Yang, Principal Investigator, Clinical Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021KYPJ202
Record Dates: First submitted 2022-02-28; First posted 2022-03-10 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Contact Lenses, Hydrophilic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): one group for contact lens
  Interventions: Device: MiSight mutifocal soft contact lens; Device: Proclear 1 Day soft contact lens

INTERVENTIONS:
Device: MiSight mutifocal soft contact lens — Subjects will wear MiSight™ multifocal soft contact lenses for 1 month.
Device: Proclear 1 Day soft contact lens — Proclear™ 1 Day soft contact lens will be worn for baseline evaluation.

SUMMARY:
The study is aimed to observe the short-term clinical performance of MiSight™ multifocal soft contact lens compared with Proclear™ 1day, including objective examination, subjective acceptability of wearers, and doctors' evaluation of the clinical manifestations of lenses.

DETAILED DESCRIPTION:
Compared with Proclear™ 1day, observe the short-term clinical performance of MiSight™ multifocal soft contact lens including objective examination, subjective acceptability of wearers, and doctors' evaluation of the clinical manifestations of lenses in 1 month.

ELIGIBILITY:
Inclusion Criteria:

* • Prior to being considered eligible to participate in this study, each subject MUST:

  1. Be between 8 and 12 years of age inclusive at the baseline examination.
  2. Have:

     1. read the Informed Assent,
     2. been given an explanation of the Informed Assent,
     3. indicated an understanding of the Informed Assent and
     4. signed the Informed Assent Form.
  3. Have their parent or legal guardian:

     1. read the Informed Consent,
     2. been given an explanation of the Informed Consent,
     3. indicated an understanding of the Informed Consent and
     4. signed the Informed Consent Form.
  4. Along with their parent or guardian, be capable of comprehending the nature of the study and be willing and able to adhere to the instructions set forth in this protocol.
  5. Along with their parent or guardian, agree to maintain the visit schedule and be able to keep all appointments as specified in the study protocol for the duration of the study.
  6. Agree to wear the assigned contact lenses for the duration of the 1-month study and to inform the study investigator if this schedule is interrupted. (Wearing time may be modified by the study staff for health reasons.)
  7. Meet the following refractive criteria determined by cycloplegic autorefraction at baseline:

     1. Spherical refractive error： between -0.75 and -4.00 D inclusive,
     2. Astigmatism: ≤-0.75 D,
     3. Anisometropia: ≤1.50D,
  8. Best-corrected visual acuity :≥0.8.

Exclusion Criteria:

* • Subjects may not be considered eligible if ANY of the following apply:

  1. Subject has regular use of ocular medications.
  2. Any systemic disease which is not suggested to wear contact lens or current use of systemic medications which may significantly affect contact lens wear, visual function, or refractive state.
  3. A history of ocular trauma or ocular surgery in the last 8 weeks.
  4. Subject has worn rigid gas permeable contact lenses in the last 6 weeks, including orthokeratology lenses.
  5. Abnormal secretion or excretion of tear fluid, infection of the tear ducts, or other recurrent ocular infections.
  6. A known allergy to fluorescein, benoxinate, proparacaine, or tropicamide.
  7. Keratoconus or an irregular cornea.
  8. Subjects who have been in a special environment such as dryness, serious dust, or volatile chemicals for a long time affect the wear of contact lenses.
  9. Strabismus, amblyopia patients, only one eye meets the admission conditions.
  10. Subjects have received any myopia control treatment.
  11. Subject is currently an active participant in another clinical study.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-07-16 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-16 (Estimated)

PRIMARY OUTCOMES:
Change in the contrast sensitivity visual function (CSF) relative to baseline at 1 month | Proclear baseline;VMisight baseline; 1 week; 1month

SECONDARY OUTCOMES:
Patients' subjective acceptability to multifocal soft contact lens | Proclear baseline; Misight baseline; 1 week; 1month
  The patients will be asked to complete questionnaires at each visit regarding vision, lens comfort, the difficulty of lens insert and removal, etc. of the multifocal contact lens.
Doctors' clinical evaluation to multifocal soft contact lens | Proclear baseline; Misight baseline; 1 week; 1month
  The doctors will be asked to complete questionnaires regarding the difficulty of fitting procedure and general impression of the multifocal contact lens.
Change in the contact lens corrected visual acuity relative to baseline | Proclear baseline;Misight baseline；1 week;1month
  Patients will wear contact lens when they are tested

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Yang, PhD, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No